CLINICAL TRIAL: NCT01709890
Title: Evaluation of a New Airway Device - the YO2(R) Catheter in Patients Under Sedation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: SZENG1.0
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Patients Undergoing Anesthesiologist-administered iv Sedation During Diagnostic/ Therapeutic Procedures
MeSH Terms: interventions — Catheters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Airway catheter during sedation
  Interventions: Device: YO2(R) catheter

INTERVENTIONS:
Device: YO2(R) catheter

SUMMARY:
Patients under sedation not uncommonly develop upper airway obstruction or other respiratory complications and no airway device is available to provide reliable maintenance of the airway at present. I believe the YO2(R)airway catheter can improve the maintenance of patent airway in most sedated patients and improve O2 delivery to the airway. In addition it may also greatly facilitate the monitoring of expired CO2, which is widely recognised as the most important monitor of adequacy of breathing, yet frequently impossible to perform satisfactorily in sedated patients at the moment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient, age >18 and <80
2. Undergoing anesthesiologist-administered sedation for diagnostic/ therapeutic procedures

Exclusion Criteria:

1. Expected procedure require access to or involve the nostrils.
2. Obesity (BMI >=30)
3. Chronic lung diseases (e.g. COPD) associated with chronic hypoxia
4. Pregnant or lactating women.
5. Known chronic liver or renal disease.
6. Mentally incapable of providing informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing anesthesiologist-administered sedation for diagnostic/ therapeutic procedures
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-12

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, The University of Hong Kong, Hong Kong, Hong Kong, China